CLINICAL TRIAL: NCT03711578
Title: An Open Label, Phase II Study to Evaluate the Efficacy and Safety of Tenalisib (RP6530), a Novel PI3K δ/γ Dual Inhibitor in Adult Patients With Relapsed/Refractory Indolent Non-Hodgkin's Lymphoma (iNHL)
Brief Title: Efficacy and Safety Study of Tenalisib (RP6530), a Novel PI3K δ/γ Dual Inhibitor in Patients With Relapsed/Refractory Indolent Non-Hodgkin's Lymphoma (iNHL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rhizen Pharmaceuticals SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP6530-1802
Record Dates: First submitted 2018-10-15; First posted 2018-10-18 (Actual); Results first posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-07

CONDITIONS: Non Hodgkin Lymphoma
Keywords: Non-Hodgkin lymphoma,; Tenalisib; RP6530
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — tenalisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tenalisib (Experimental): Participants receive Tenalisib 800 mg BID in 28-Days Cycle for 8 Cycles
  Interventions: Drug: Tenalisib,

INTERVENTIONS:
Drug: Tenalisib, — BID, Orally
  Other Names: RP6530

SUMMARY:
To assess the anti-tumor activity and safety of Tenalisib in patients with relapsed/refractory indolent Non-Hodgkin's Lymphoma (iNHL),

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed diagnosis of indolent B-cell NHL, with histological subtype limited to:

   1. Follicular lymphoma (FL) G1, G2, or G3a
   2. Marginal zone lymphoma (MZL) (splenic, nodal, or extra-nodal)
   3. Lymphoplasmacytic lymphoma/Waldenstrom macroglobulinemia (LPL/WM)
   4. Small lymphocytic lymphoma (SLL) with absolute lymphocyte count <5 x10^9/L at the time of diagnosis and at study entry.
2. Relapsed or refractory after ≥ 2 prior lines of therapy (refractory defined as not responding to a standard regimen or progressing within 6 months of the last course of a standard regimen). Patients must have received rituximab and alkylating agents.
3. Patients must have at least one bi-dimensionally measurable lesion (that has not been previously irradiated) with the longest diameter ≥ 1.5 cm.
4. Male or female patients > 18 years of age.
5. ECOG performance status ≤ 2.
6. Life expectancy of at least 3 months.
7. Adequate bone marrow, liver, and renal function as assessed by the following laboratory requirements conducted within 7 days before starting study treatment:

   1. Hemoglobin ≥ 9 g/dl
   2. Absolute neutrophil count (ANC) ≥ 1 x 10^9/L
   3. Platelets ≥50 x 10^9/L (patient without BM involvement) and 30 x 10^9/L (patient with BM involvement)
   4. Total bilirubin ≤1.5 times the upper limit of normal (ULN)
   5. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 x ULN if known liver involvement
   6. Creatinine ≤ 1.5 mg/dL OR calculated creatinine clearance ≥ 50 mL/min (as calculated by the Cockcroft-Gault method)
8. Use of an effective means of contraception for female patients of child-bearing potential, and all male partners.
9. Willingness and ability to comply with trial and follow-up procedures, give written informed consent.

Exclusion Criteria:

1. FL grade 3b or transformed disease or CLL
2. Cancer therapy within 3 weeks (21 days) or 5 half-lives (whichever is shorter) prior to C1D1. Corticosteroids (prednisone or equivalent) at a dose of < 20 mg daily are allowed. Corticosteroid should be stabilized for at least 1 week prior to C1D1
3. Auto-SCT within 3 months from C1D1 (patients must not have active graft versus- host disease)
4. History of having received an Allo-SCT
5. Active hepatitis B or C infection
6. Known history of human immunodeficiency virus (HIV) infection
7. Evidence of ongoing severe systemic bacterial, fungal or viral infection
8. Known primary central nervous system lymphoma or any preexisting neurologic manifestations
9. Known history of drug-induced liver injury, alcoholic liver disease, primary biliary cirrhosis, ongoing extrahepatic obstruction caused by stones, cirrhosis of the liver or portal hypertension;
10. Prior exposure to drug that specifically inhibits PI3K
11. Pregnancy or lactation
12. Myeloid growth factors or red blood cells/ platelet transfusion within 14 days prior to C1D1
13. Drug administration within 1 week prior to C1D1

    1. Strong inhibitors or inducers of CYP3A4, CYP2C9, including grapefruit products, herbal supplements and drugs
    2. Substrates of CYP3A4 enzyme with a narrow therapeutic range

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-11-25 (Actual); Primary Completion 2020-06-16 (Actual); Study Completion 2020-10-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (8):
  - Clearview Cancer Institute, Huntsville, Alabama
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Florida cancer specialists & Research Institute, Florida City, Florida
  - Florida Cancer Specialist/ South, Fort Myers, Florida
  - Florida Cancer Specialists/North, St. Petersburg, Florida
  - HCA Midwest Health Kansas City, Kansas City, Missouri
  - Tennessee Oncology, Chattanooga, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
- Australia (4):
  - Blacktown Hospital, Blacktown Cancer and Haematology Center, Blacktown, New South Wales
  - Brisbane Clinic for Lymphoma, Myeloma and Leukaemia,, Greenslopes, Queensland
  - John Flynn Private Hospital,, Tugun, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tenalisib
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tenalisib
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 11
Age, Continuous [Median (Full Range); unit: years] | 66.575 [46.95 to 83.54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11
  Australia | 9

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as sum of CR and PR rates and will be assessed according to the Lugano Classification for initial evaluation, staging, and response assessment of Non-Hodgkin lymphoma. (Cheson-2014)
Time Frame: 7 months
Population: Patients who received at least 1 dose of study medication and provided at least 1 post-baseline efficacy assessment
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Tenalisib
Number analyzed (Participants) | 19
Percent of participants | 5.3 [0.13 to 26.03]

2. Primary Outcome: Complete Response Rate
Description: CR rate will be assessed according to the Lugano Classification for initial evaluation, staging, and response assessment of non-Hodgkin lymphoma.
Time Frame: 7 months
Population: Patients who received at least 1 dose of study medication and provided at least 1 post-baseline efficacy assessment
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Tenalisib
Number analyzed (Participants) | 19
Percent of participants | 0.00 [0 to 17.65]

3. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time of the first dose of Tenalisib to disease progression or death.
Time Frame: From date of first dose of tenalisib until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 7 months
Population: Patients who received at least 1 dose of study medication and provide at least 1 post-baseline efficacy assessment
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Tenalisib
Number analyzed (Participants) | 19
days | 113 [57 to 275]

4. Primary Outcome: Duration of Response (DoR)
Description: DoR is measured from the initial response to disease progression or death
Time Frame: 7 months
Population: Patients who received at least 1 dose of study medication and provide at least 1 post-baseline efficacy assessment
Measure: Number; unit: days
Arm/Group | Tenalisib
Number analyzed (Participants) | 19
days | 0

5. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events as Assessed by CTCAE v4.0
Description: Safety and tolerability of Tenalisib
Time Frame: 8 months
Population: Patients who received at least 1 dose of study medication
Measure: Number; unit: participants
Arm/Group | Tenalisib
Number analyzed (Participants) | 20
participants | 18

ADVERSE EVENTS:
Time Frame: 8 months
Description: Summary of Treatment-Emergent Adverse Events-(Causality All). Patients were monitored for adverse events and both related and as well as non-related adverse events were captured during the study. All adverse events (irrespective of causality) are reported here.
Arm/Group | Tenalisib
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 3/20
Other Adverse Events (participants affected / at risk) | 13/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tenalisib (N=20)
Pyrexia (General disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tenalisib (N=20)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 5 (5)
Chills (General disorders) | 1 (2)
Pyrexia (General disorders) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 2 (2)
Neutrophil Count Decreased (Investigations) | 2 (3)
Alanine aminotransferase increased (Investigations) | 1 (3)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (5)
Dysgeusia (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (3)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Eructation (Gastrointestinal disorders) | 1 (1)
Influenza like illness (General disorders) | 1 (1)
Allergy to arthropod bite (Immune system disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Escherichia urinary tract infection (Infections and infestations) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1)
Serratia infection (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (2)
Platelet count decreased (Investigations) | 1 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neurological symptoms (Nervous system disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Nocturia (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Rash generalized (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-12-04): https://cdn.clinicaltrials.gov/large-docs/78/NCT03711578/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-07): https://cdn.clinicaltrials.gov/large-docs/78/NCT03711578/SAP_002.pdf